CLINICAL TRIAL: NCT05293769
Title: Reliability of a Food Frequency Questionnaire in the Assessment of Dietary Intake Including FODMAPs (Fermentable Oligosaccharides, Disaccharides, Monosaccharides and Polyols) in Different Populations, and Relationship With IBS (Inflammatory Bowel Syndrome) Symptoms and the Degree of Self-assessed Physical Activity
Brief Title: Reliability of a Food Frequency Questionnaire in the Assessment of Dietary Intake Including FODMAPs in Different Populations, and Relationship With IBS Symptoms and the Degree of Self-assessed Physical Activity
Status: Recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: FaST
Record Dates: First submitted 2021-10-27; First posted 2022-03-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBS - arm
  Interventions: Other: questionnaire
- healthy - arm
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — questionnaire will be filled in by all participants

SUMMARY:
During an online assessment participants will fill in questionnaires evaluating demographic data, psychological variables, the degree of self-assessed physical activity and symptoms of irritable bowel. Dietary intake will be assessed by a newly developed food frequency questionnaire (FFQ) and a 4 days food diary. In order to validate the FFQ in different populations, participants will be recruited from university students, staff of UZ Brussel and VUB, and from the community by advertisement (including social media). IBS patients will be recruited from the gastro-enterology outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years;
* Provide written informed consent;
* Living in Belgium

Exclusion Criteria:

* Diet < 8 weeks prior to participation;
* Known or suspected eating disorder;
* Major psychiatric disorder;
* Known gastro-intestinal disease (IBS is allowed);
* Any malignancy in the past 3 years (basocellular carcinoma is allowed);
* Chemotherapy in the past 6 months;
* Infectious gastro-enteritis in the past 6 months (infectious gastro-enteritis defined as the concurrent presence of one of the following signs during 2 or more consecutive days: fever, vomiting, sudden onset of diarrhea, hospitalization because of these symptoms);
* Previous abdominal surgery (appendectomy and cholecystectomy are allowed);
* Alcohol abuse defined as > 14 U per week;
* Use of illicit drugs;
* Intake of drugs with known major gastro-intestinal side effects.
* Initiation of neuromodulators less than 3 months before participation. Neuromodulators are allowed when taken at a stable dose for at least 3 months;
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy subjects, IBS patients
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
To validate the newly developed food frequency questionnaire against the standard 4-day food diary across different populations | 2 years

SECONDARY OUTCOMES:
Comparison of dietary and FODMAP intake in IBS vs. non-IBS patients in different populations | 2 years
  differences in number and type of FODMAP intake between groups
Comparison of the degree of physical activity in IBS vs. non-IBS patients in different populations | 2 years
  differences and correlation of IPAQ (International Physical Activity Questionnaire) scores between groups, IPAQ evaluates the level of physical activity. Scoring a HIGH level of physical activity on the IPAQ means your physical activity levels equate to approximately one hour of activity per day or more
Comparison of the degree of physical activity and IBS symptom severity in different populations | 2 years
  differences and correlation of IPAQ scores between groups; IPAQ evaluates the level of physical activity. Scoring a HIGH level of physical activity on the IPAQ means your physical activity levels equate to approximately one hour of activity per day or more

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No